CLINICAL TRIAL: NCT05020015
Title: A Phase 2, Open-label, Multicenter Study of the Safety and Efficacy of TAK-007 in Adult Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Brief Title: A Study of TAK-007 in Adults With Relapsed or Refractory (r/r) B-cell Non-Hodgkin Lymphoma (NHL)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TAK-007-2001; 2021-002086-18 (EudraCT Number)
Record Dates: First submitted 2021-08-20; First posted 2021-08-25 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Relapsed or Refractory (r/r) B-cell Non-Hodgkin Lymphoma (NHL)
Keywords: Drug Therapy; Chimeric antigen receptor; Natural killer cells; Cell therapy; Allogeneic
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: This study has 2 Parts: Part 1 is composed of dose escalation followed by dose expansion and Part 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells (Experimental): Participants received lymphodepleting chemotherapy per day intravenously (IV) for 3 days followed by TAK-007 200×10^6 anti-CD19 chimeric antigen receptor (CD19-CAR+) viable NK cells, single-dose, IV infusion, once on Day 0.
  Interventions: Biological: TAK-007; Drug: Chemotherapy Agents
- Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells (Experimental): Participants received lymphodepleting chemotherapy per day IV for 3 days followed by TAK-007 - 800×10^6 CD19-CAR+ viable NK cells, single-dose, IV infusion, once on Day 0.
  Interventions: Biological: TAK-007; Drug: Chemotherapy Agents
- Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells (Experimental): Participants with r/r LBCL received lymphodepleting chemotherapy per day IV for 3 days followed by TAK-007 at the dose level selected based on the dose escalation part (800×10^6 CD19-CAR+ viable NK cells), as a single-dose, IV infusion, once on Day 0 to determine recommended phase 2 dose (RP2D).
  Interventions: Biological: TAK-007; Drug: Chemotherapy Agents
- Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells (Experimental): Participants with r/r iNHL received lymphodepleting chemotherapy per day IV for 3 days followed by TAK-007 at the dose level(s) selected based on the dose escalation part (800×10^6 CD19-CAR+ viable NK cells), as a single-dose, IV infusion, once on Day 0 to determine RP2D.
  Interventions: Biological: TAK-007; Drug: Chemotherapy Agents

INTERVENTIONS:
Biological: TAK-007 — TAK-007 intravenous injection.
Drug: Chemotherapy Agents — Fludarabine and cyclophosphamide as per standard of care.

SUMMARY:
This study has 2 parts.

The main aim of Part 1 is to check for side effects from TAK-007 in adults with relapsed or refractory (r/r) B-cell Non-Hodgkin Lymphoma (NHL),

The main aim of Part 2 is to learn whether lymphoma disease responds to treatment with TAK-007 in adults with r/r B-cell NHL or iNHL.

Participants will receive 3 days of chemotherapy to reduce a type of white blood cells called lymphocytes, in the blood. This is called lymphodepleting chemotherapy (LDC) or lymphodepletion. After LDC, patients will receive a single injection of TAK-007 or three weekly injections of TAK-007 (multi-dose injection). After this, participants will regularly visit the clinic for check-ups.

DETAILED DESCRIPTION:
The product being tested in this study is called TAK-007. TAK-007 is being tested to evaluate the safety and tolerability in adult participants with r/r B-cell NHL. The study will include 2 parts: Part 1 (Dose escalation and dose expansion) and Part 2.

The study will enroll approximately 265 participants.

In Part 1, dose escalation cohorts' participants will receive TAK-007 as follows:

Part 1 dose escalation:

* Part 1: Dose escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK (Natural Killer) Cells (±30%)
* Part 1: Dose escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells (±25%)

In Part 1 dose expansion phase, separate expansion cohorts for LBCL and iNHL (Cohorts 1A [LBCL 3L+] and 2A [iNHL 3L+]) and two additional dose expansion cohorts with a multi-dose regimen will be added (i.e., Cohort 1B and 1C) to evaluate more than 1 doses of TAK-007 after a 3-day regimen of lymphodepleting chemotherapy.

Part 1 dose expansion cohorts' participants will receive TAK-007 as follows:

* Part 1: Dose expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells on Day 0 of the study.
* Part 1: Dose expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells on Day 0 of the study.

Based on the data in Part 1, a single TAK-007 dose level will be selected by the sponsor and investigators as the recommended phase 2 dose (RP2D).

Once RP2D is determined, participants will be enrolled in Part 2 of the study in the following cohorts:

* Cohort 1: TAK-007 (LBCL)
* Cohort 2: TAK-007 (iNHL)

This multi-center trial will be conducted worldwide. Part 1 of the study will be conducted in the US, and Part 2 will be conducted worldwide. The overall time to participate in this study is 5 years. Participants will make multiple visits to the clinic and will enroll in a separate, long-term, follow-up study for continued safety assessments for up to 15 years after TAK-007 administration.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who have a life expectancy ≥12 weeks.
2. Participants who have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
3. Participants with a diagnosis of previously treated r/r histologically proven Cluster of Differentiation (CD)19 expressing disease of the following types:

   a. LBCL, including the following subtypes defined by the World Health Organization (WHO): i. Diffuse large B-cell lymphoma (DLBCL) not otherwise specified (NOS). ii. High-grade B-cell lymphoma (HGBL) with MYC and BCL2 and/or BCL6 rearrangement iii. HGBL NOS without translocations. iv. DLBCL arising from iNHL including follicular lymphoma (FL) or marginal zone lymphoma (MZL).

   v. T-cell/histiocyte-rich LBCL. vi. DLBCL associated with chronic inflammation. vii. Epstein-Barr virus-positive DLBCL-NOS. viii. Primary cutaneous DLBCL, leg type. ix. Primary mediastinal large B-cell lymphoma (PMBCL). x. FL Grade 3B. b. iNHL, including the following subtypes defined by the WHO: i. FL Grades 1, 2, 3A. ii. MZL (nodal, extranodal, and splenic).
4. Participants who have measurable disease, defined as at least 1 lesion per the Lugano classification. Lesions situated in a previously irradiated area are considered measurable if radiographic progression has been documented in such lesions following completion of radiation therapy. LBCL should have positron emission tomography (PET) -positive disease per the Lugano classification.
5. Participants who have r/r LBCL or r/r iNHL after ≥2 prior lines of systemic therapy: (Expansion Cohorts 1A and 1B [LBCL 3L+], and 2A [iNHL 3L +]) or r/r LBCL after 1 prior line of systemic therapy (Expansion Cohort 1C [LBCL 2L]):

   1. Participants with r/r LBCL must have received an anti-CD20 monoclonal antibody (mAb) and an anthracycline containing chemotherapy regimen and failed or be ineligible for high-dose chemotherapy and autologous stem cell transplantation (ASCT).
   2. Participants with iNHL must have received an anti-CD20 mAb and an alkylating agent (eg, bendamustine or cyclophosphamide).
   3. Preinduction salvage chemotherapy and ASCT should be considered 1 line of therapy.
   4. Any consolidation/maintenance therapy after a chemotherapy regimen (without intervening relapse) should be considered 1 line of therapy with the preceding combination therapy. Maintenance antibody therapy should not be considered a line of therapy.
   5. Single-agent anti-CD20 mAb therapy should not be considered a line of therapy.
   6. Bridging chemotherapy given just prior to CAR-T cell therapy treatment should be considered one line of therapy together with cell therapy.
   7. Participants who have received prior CD19-targeting CAR-T cell therapy must have achieved at least a partial response to the most recent CD19-targeting CAR-T cell therapy.
   8. Participants with 1 prior line of therapy in Part 1 Cohort 1C must have either:

      * refractory disease to first-line chemoimmunotherapy or relapse within 12 months of first-line chemoimmunotherapy OR
      * relapsed or refractory disease and be ineligible for intensive chemoimmunotherapy and/or high-dose chemotherapy followed by ASCT due to comorbidities and/or age.
6. Participants who have adequate bone marrow function defined as follows:

   1. Absolute neutrophil count >500/μL.
   2. Platelet count of >50,000/μL at screening. Participants with transfusion-dependent thrombocytopenia are excluded.
7. Participants who have adequate renal, hepatic, cardiac, and pulmonary function as defined in the study protocol:

   1. Estimated glomerular filtration rate (GFR; Modification of Diet in Renal Disease equation [MDRD]) ≥30 mL/min.
   2. Serum alanine aminotransferase/aspartate aminotransferase ≤5 times the upper limit of normal range (ULN), as long as participant is asymptomatic.
   3. Total bilirubin ≤2 mg/dL. Participants with Gilbert's syndrome may have a bilirubin level >2 × ULN, per discussion between the investigator and the medical monitor.
   4. Left ventricular ejection fraction (LVEF) ≥40% as determined by an echocardiogram (ECHO) or multigated acquisition (MUGA) scan performed within 1 month of determination of eligibility.
   5. No evidence of clinically relevant pericardial effusion, and no acute clinically significant electrocardiogram (ECG) findings.
   6. Absence of Grade ≥2 pleural effusion. Grade 1 stable pleural effusions are allowed.
   7. Baseline oxygen saturation >92% on room air.
8. Participants are required to consent to provide either sufficient archived formalin-fixed paraffin embedded (at least 10 unstained slides, ideally 20 unstained slides) or fresh tumor tissue obtained after the last relapse (see laboratory manual for details). Exception may be granted by sponsor medical monitor per discussion with investigator.

Exclusion Criteria:

1. Participants with total body weight of <40 kg.
2. Participants with primary or secondary central nervous system (CNS) involvement by lymphoma. Participants with a history of secondary CNS involvement by lymphoma without evidence of CNS involvement at screening may be included.
3. Participants with Burkitt lymphoma, mantle cell lymphoma, lymphoplasmocytic lymphoma, or transformation from CLL/small lymphocytic lymphoma (Richter transformation).
4. Participants with a history of malignancy other than nonmelanoma skin cancer, carcinoma in situ (eg, cervix, bladder, breast), low-grade tumors deemed to be cured and not treated with systemic therapy (eg, by gastro-endoscopy curatively removed gastric cancer) or unless disease free for ≥3 years at screening.
5. Participants who have undergone autologous or allogeneic transplant or Chimeric antigen receptor T cells (CAR-T) or Chimeric antigen receptor Natural Killer cells (CAR-NK) therapy within 3 months of planned enrollment. Participants after allogeneic transplant have to be off systemic immunosuppressive therapy and without the evidence of clinically relevant acute or chronic graft-versus-host disease (GvHD) at the time of enrollment.
6. Treatment with any investigational products or any systemic anticancer treatment within 14 days or 2 half-lives of the treatment (whichever is longer) before conditioning therapy. For rituximab, a half-life of 22 days should be considered.
7. Participants with active infection, including fungal, bacterial, viral, or other infection that is uncontrolled or requires IV antimicrobials for management within 3 days before enrollment.
8. Participants with a history or presence of active or clinically relevant CNS disorder, such as seizure, encephalopathy, cerebrovascular ischemia/hemorrhage, severe dementia, cerebellar disease, or any autoimmune disease with CNS involvement. For CNS disorders that recover or are in remission, participants without recurrence within 2 years of planned study enrollment may be included.
9. Participants with any of the following within 6 months of enrollment: myocardial infarction, cardiac angioplasty or stenting, unstable angina, symptomatic congestive heart failure (ie, New York Heart Association Class II or greater), clinically significant arrythmia (including uncontrolled atrial fibrillation), or any other clinically significant cardiac disease.
10. Participants who have received a live vaccine ≤6 weeks before the start of the conditioning regime.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2024-06-16 (Actual); Study Completion 2038-12-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (15):
- United States (15):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - MedStar Georgetown University Medical Center, Washington D.C., District of Columbia
  - Sylvester Comprehensive Cancer Center University of Miami Hospitals and Clinics, Miami, Florida
  - Northside Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - DUHS Duke Blood Cancer Center, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University Sidney Kimmer Cancer Center, Clinical Research Organization, Philadelphia, Pennsylvania
  - Saint Davids South Austin Medical Center, Austin, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/612723b3ca0ce2002ab9e667

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the investigative sites in the United States (US) from 12 November 2021 to 01 July 2024 (data cut off). The study is ongoing.
Pre-assignment Details: Participants with relapsed or refractory (r/r) B-cell non-Hodgkin lymphoma (NHL), including large B-cell lymphoma (LBCL) participants who have failed ≥2 prior systemic therapies (i.e., third or higher line [3L+] treatment) and indolent non-Hodgkin lymphoma (iNHL) participants who have failed ≥2 prior systemic therapies (3L+) were included in this study. Part 2 will no longer be initiated and conducted as per the latest protocol amendment for this study.
Period: Overall Study
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Started | 3 | 6 | 11 | 7
Completed | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 11 | 7
Not completed — Ongoing on study | 1 | 3 | 4 | 7
Not completed — Death | 2 | 3 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Reason Not Specified | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) set included all enrolled participants in the TAK-007 study.
Groups:
- Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells: Participants received lymphodepleting chemotherapy per day IV for 3 days followed by TAK-007 -200×10^6 CD19-CAR+ viable NK cells, single-dose, IV infusion, once on Day 0.
- Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells: Participants with r/r LBCL received lymphodepleting chemotherapy per day IV for 3 days followed by TAK-007 at the dose level selected based on the dose escalation part (800×10^6 CD19-CAR+ viable NK cells), as a single-dose, IV infusion, once on Day 0 to determine RP2D.
- Total: Total of all reporting groups
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Total
Number analyzed (Participants) | 3 | 6 | 11 | 7 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (5.29) | 61.5 (9.01) | 63.2 (10.87) | 66.6 (10.58) | 63.7 (9.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4 | 8
  Male | 2 | 5 | 9 | 3 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 6 | 10 | 6 | 25
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 3 | 6 | 8 | 7 | 24
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a study intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the study intervention or medicinal product.
Time Frame: Up to 24 months
Population: Safety Analysis Set included all participants who received TAK-007 administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 3 | 6 | 10 | 7
Participants | 3 | 6 | 10 | 7

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Laboratory Parameters
Description: Laboratory parameters included hematology, clinical chemistry, serum immunoglobulin and urinalysis tests.
Time Frame: Up to 24 months
Population: Safety Analysis Set included all participants who received TAK-007 administration.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 200×10^6 or 800×10^6 CD19-CAR+ Viable NK Cells: Participants with r/r LBCL received lymphodepleting chemotherapy per day IV for 3 days followed by TAK-007 at the dose level selected based on the dose escalation part (800×10^6 CD19-CAR+ viable NK cells), as a single-dose, IV infusion, once on Day 0 to determine RP2D.
- Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 200×10^6 or 800×10^6 CD19-CAR+ Viable NK Cells: Participants with r/r iNHL received lymphodepleting chemotherapy per day IV for 3 days followed by TAK-007 at the dose level(s) selected based on the dose escalation part(200×10^6 or 800×10^6 CD19-CAR+ viable NK cells), as a single-dose, IV infusion, once on Day 0 to determine RP2D.
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 200×10^6 or 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 200×10^6 or 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 3 | 6 | 10 | 7
Participants
  Hemoglobin | 2 | 5 | 7 | 2
  Leukocytes | 3 | 5 | 10 | 7
  Lymphocytes | 3 | 6 | 7 | 7
  Neutrophils | 3 | 6 | 10 | 7
  Platelets | 2 | 3 | 4 | 3
  Alanine aminotransferase (ALT) | 0 | 0 | 1 | 0
  Albumin | 1 | 3 | 2 | 1
  Aspartate aminotransferase (AST) | 0 | 0 | 1 | 0
  Bilirubin | 0 | 1 | 0 | 0
  Creatinine | 0 | 1 | 2 | 1
  Estimated glomerular filtration rate (GFR) | 1 | 2 | 3 | 2
  Potassium | 0 | 0 | 1 | 0
  Sodium | 1 | 1 | 0 | 1
  Immunoglobulin G | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Notable Changes in Vital Signs
Description: Vital signs included body temperature (oral or tympanic measurement), sitting blood pressure (after the participant had rested for at least 5 minutes), and pulse rate (beats per minute [bpm]).
Time Frame: Up to 24 months
Population: Safety Analysis Set included all participants who received TAK-007 administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 3 | 6 | 10 | 7
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: ORR Per Investigator
Description: ORR is defined as the percentage of participants with CR or PR as best response to treatment, determined by the investigator per the Lugano 2014 criteria after TAK-007 administration. CR is defined as percentage of participants with target nodes/nodal masses must regress to ≤1.5 cm in the longest transverse diameter of all lesions and no extralymphatic sites of disease. PR is defined as ≥50% decrease in sum of the product of the perpendicular diameters of up to 6 target measurable nodes and extranodal sites; absent/normal, regressed, but no increase in nonmeasured lesion; Spleen must have regressed by >50% in length beyond normal.
Time Frame: Up to 24 months
Population: Modified Intent-to-Treat (mITT) set included all participants who received TAK-007 administration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 3 | 6 | 10 | 7
percentage of participants | 0 [0.0 to 70.8] | 50.0 [11.8 to 88.2] | 50.0 [18.7 to 81.3] | 85.7 [42.1 to 99.6]

5. Secondary Outcome: Complete Response (CR) Per Investigator
Description: CR is defined per Lugano 2014 criteria as percentage of participants with target nodes/nodal masses must regress to ≤1.5 cm in the longest transverse diameter of all lesions and no extralymphatic sites of disease.
Time Frame: Up to 24 months
Population: mITT set included all participants who received TAK-007 administration.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 3 | 6 | 10 | 7
percentage of participants | 0 [0.0 to 70.8] | 33.3 [4.3 to 77.7] | 20.0 [2.5 to 55.6] | 57.1 [18.4 to 90.1]

6. Secondary Outcome: Duration of Response (DOR) Per Investigator
Description: DOR is defined only for participants who experienced objective response (complete response or partial response) and is the time from the date of first documented objective response to the date of first documented disease progression or death, whichever comes first. Participants not meeting the criteria for progression or death will be censored at the last disease assessment.
Time Frame: Up to 24 months
Population: mITT set included all participants who received TAK-007 administration. Overall number of participants analyzed is the number of participants with events.
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 0 | 3 | 5 | 6
months |  | 4.9 [2.5 to 8.0] | 2.4 [0.0 to 4.5] | 4.9 [1.8 to 7.9]

7. Secondary Outcome: Progression-free Survival (PFS) Per Investigator
Description: Progression-free survival is defined as the time from TAK-007 administration to the date of disease progression or death from any cause, whichever comes first. Participants who do not have disease progression or die were censored at the last disease assessment. Participants who do not have postbaseline disease assessment prior to new anticancer therapy (excluding SCT) in the absence of death were censored at the dosing date of TAK-007.
Time Frame: Up to 24 months
Population: mITT set included all participants who received TAK-007 administration.
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 3 | 6 | 10 | 7
months | 0.95 [0.85 to 1.02] | 2.23 [0.95 to 9.00] | 2.00 [0.03 to 5.55] | 5.62 [2.83 to 8.77]

8. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from TAK-007 administration to the date of death. Participants who did not die were censored at the last contact date.
Time Frame: Up to 24 months
Population: mITT set included all participants who received TAK-007 administration.
Measure: Median (Full Range); unit: months
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 3 | 6 | 10 | 7
months | 8.9 [1.7 to 20.3] | NA [1.5 to 18.3] — Median was not estimable due to insufficient number of participants with events. | 8.4 [0.9 to 11.2] | NA [6.0 to 13.8] — Median was not estimable due to insufficient number of participants with events.

9. Secondary Outcome: Cmax - Maximum Observed Blood Concentration of TAK-007
Description: The unit of measure 'copies per microgram' indicates copies of TAK-007 transgene per micrograms of genomic deoxyribonucleic acid (DNA).
Time Frame: At 1 hour (±15 minutes) predose and postdose (Day 0) and once on Days 1, 3, 7, 10, 14, 21, 28/Month 1, Months 2, 3, 4, 6, 9, 12, 18, 24
Population: Cellular kinetic (CK) analysis set included all participants who received TAK-007 administration and had at least 1 plasma sample obtained and analyzed. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Mean (Standard Deviation); unit: copies per microgram (µg)
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 2 | 6 | 6 | 8
copies per microgram (µg) | 1140 (299) | 4730 (8500) | 6540 (4510) | 15800 (28500)

10. Secondary Outcome: Tmax - Time of First Occurrence of Cmax of TAK-007
Time Frame: as for outcome 9
Population: CK analysis set included all participants who received TAK-007 administration and had at least 1 plasma sample obtained and analyzed. Overall number of participants analyzed is the number of participants with data available for analysis.
Measure: Median (Full Range); unit: days
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 2 | 6 | 6 | 8
days | 0.05 [0.04 to 0.05] | 0.31 [0.04 to 15.07] | 0.04 [0.04 to 0.05] | 0.05 [0.04 to 91.91]

11. Secondary Outcome: Tlast - Time of Last Measurable Concentration Above the Lower Limit of Quantitation of TAK-007
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Median (Full Range); unit: days
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 2 | 6 | 6 | 8
days | 0.05 [0.04 to 0.05] | 5.39 [0.05 to 15.07] | 0.05 [0.04 to 13.83] | 6.87 [0.04 to 176.98]

12. Secondary Outcome: AUClast - Area Under the Concentration-time Curve From Time 0 to Time of the Last Quantifiable Concentration of TAK-007
Description: The unit of measure 'day*copies/µg' indicates day*copies of TAK-007 transgene per µg of genomic DNA.
Time Frame: as for outcome 9
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: day*copies/µg
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 2 | 6 | 6 | 8
day*copies/µg | 25.9 (8.41) | 1100 (1130) | 8330 (12800) | 825000 (2240000)

13. Secondary Outcome: Concentration of Interleukin (IL)-15 and Other Soluble Immune Factors in Plasma Over Time
Description: Concentration of IL-15 and soluble immune factors (eg, Interferon (IFN)-gamma (γ) and IL-6) in plasma over time were reported.
Time Frame: Baseline, pre-dose (Day 0) and post-dose at Days 1, 7, 14, 21, 28 and Months 2,3,4,6,9,12
Population: Pharmacodynamic Analysis Set included all participants from the safety analysis set who had a baseline and at least 1 postbaseline sample assessment. Number analyzed is the number of participants with data available for analysis at the specified timepoints.
Measure: Mean (Standard Deviation); unit: picograms per milliter (pg/mL)
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 3 | 5 | 10 | 7
picograms per milliter (pg/mL)
  IL-15: Baseline | 3.855 (1.0355) | 3.991 (1.6857) | 5.059 (3.7114) | 2.802 (1.0243)
  IL-15: Pre-dose: number analyzed (Participants) | 3 | 5 | 10 | 6
  IL-15: Pre-dose | 33.737 (8.6072) | 56.035 (23.7989) | 34.547 (14.5419) | 44.125 (29.8318)
  IL-15: Day 1 | 38.175 (12.2965) | 51.992 (26.7839) | 31.473 (14.1248) | 38.546 (26.6800)
  IL-15: Day 7: number analyzed (Participants) | 3 | 4 | 9 | 6
  IL-15: Day 7 | 18.288 (8.7229) | 18.364 (9.4926) | 15.775 (9.6798) | 13.434 (6.9273)
  IL-15: Day 14 | 10.342 (0.8935) | 9.384 (3.2634) | 13.592 (8.2004) | 10.707 (3.8889)
  IL-15: Day 21 | 7.915 (1.8965) | 7.734 (3.4047) | 9.900 (6.4358) | 6.176 (2.6925)
  IL-15: Day 28: number analyzed (Participants) | 1 | 5 | 8 | 6
  IL-15: Day 28 | 6.843 (NA) — Standard Deviation (SD) was not estimable for a single participant. | 12.127 (10.5958) | 5.200 (2.0747) | 4.540 (2.6362)
  IL-15: Month 2: number analyzed (Participants) | 0 | 2 | 5 | 7
  IL-15: Month 2 |  | 8.975 (6.6271) | 4.242 (1.9915) | 2.867 (0.5611)
  IL-15: Month 3: number analyzed (Participants) | 0 | 1 | 3 | 7
  IL-15: Month 3 |  | 2.669 (NA) — SD was not estimable for a single participant. | 4.149 (1.9754) | 2.409 (0.5595)
  IL-15: Month 4: number analyzed (Participants) | 0 | 1 | 1 | 4
  IL-15: Month 4 |  | 2.543 (NA) — SD was not estimable for a single participant. | 3.820 (NA) — SD was not estimable for a single participant. | 2.100 (0.0263)
  IL-15: Month 6: number analyzed (Participants) | 0 | 1 | 1 | 5
  IL-15: Month 6 |  | 2.667 (NA) — SD was not estimable for a single participant. | 2.575 (NA) — SD was not estimable for a single participant. | 2.039 (0.3939)
  IL-15: Month 9: number analyzed (Participants) | 0 | 0 | 0 | 2
  IL-15: Month 9 |  |  |  | 2.685 (0.9093)
  IL-15: Month 12: number analyzed (Participants) | 0 | 0 | 0 | 1
  IL-15: Month 12 |  |  |  | 2.613 (NA) — SD was not estimable for a single participant.
  IFN-g: Baseline | 31.558 (24.9063) | 22.738 (9.8730) | 51.761 (120.7897) | 37.396 (52.8148)
  IFN-g: Pre-dose: number analyzed (Participants) | 3 | 5 | 10 | 6
  IFN-g: Pre-dose | 41.471 (39.3018) | 35.890 (36.3154) | 24.548 (44.4643) | 96.015 (150.1385)
  IFN-g: Day 1 | 81.089 (102.7746) | 50.657 (42.5779) | 26.694 (35.6445) | 172.001 (347.0450)
  IFN-g: Day 7: number analyzed (Participants) | 3 | 4 | 9 | 6
  IFN-g: Day 7 | 56.935 (68.4453) | 44.602 (15.4926) | 31.201 (61.1626) | 29.970 (20.1722)
  IFN-g: Day 14 | 12.037 (11.1691) | 70.825 (70.1581) | 28.009 (30.1577) | 155.058 (233.9229)
  IFN-g: Day 21 | 14.645 (0.4215) | 57.785 (76.0284) | 86.566 (122.4368) | 51.144 (46.2887)
  IFN-g: Day 28: number analyzed (Participants) | 2 | 5 | 8 | 6
  IFN-g: Day 28 | 10.618 (6.7349) | 36.489 (54.2244) | 35.749 (30.4532) | 57.836 (34.8662)
  IFN-g: Month 2: number analyzed (Participants) | 0 | 2 | 5 | 7
  IFN-g: Month 2 |  | 29.038 (15.3845) | 27.540 (18.7882) | 26.493 (28.8072)
  IFN-g: Month 3: number analyzed (Participants) | 0 | 1 | 3 | 7
  IFN-g: Month 3 |  | 10.806 (NA) — SD was not estimable for a single participant. | 11.565 (7.1666) | 9.016 (5.5790)
  IFN-g: Month 4: number analyzed (Participants) | 0 | 1 | 1 | 4
  IFN-g: Month 4 |  | 11.649 (NA) — SD was not estimable for a single participant. | 13.138 (NA) — SD was not estimable for a single participant. | 11.405 (4.1568)
  IFN-g: Month 6: number analyzed (Participants) | 0 | 1 | 1 | 5
  IFN-g: Month 6 |  | 35.829 (NA) — SD was not estimable for a single participant. | 8.848 (NA) — SD was not estimable for a single participant. | 15.160 (11.9336)
  IFN-g: Month 9: number analyzed (Participants) | 0 | 0 | 0 | 2
  IFN-g: Month 9 |  |  |  | 8.254 (3.8536)
  IFN-g: Month 12: number analyzed (Participants) | 0 | 0 | 0 | 1
  IFN-g: Month 12 |  |  |  | 12.077 (NA) — SD was not estimable for a single participant.
  IL-6: Baseline | 4.289 (4.8094) | 17.169 (17.2708) | 3.453 (3.1142) | 4.129 (7.7186)
  IL-6: Pre-dose: number analyzed (Participants) | 3 | 5 | 10 | 6
  IL-6: Pre-dose | 4.814 (4.5419) | 14.454 (13.7658) | 2.309 (2.0751) | 6.776 (8.2117)
  IL-6: Day 1 | 8.993 (9.6177) | 17.015 (16.4689) | 2.295 (2.4267) | 158.548 (406.9127)
  IL-6: Day 7: number analyzed (Participants) | 3 | 4 | 9 | 6
  IL-6: Day 7 | 9.236 (12.7713) | 70.663 (106.7221) | 3.169 (3.8668) | 19.255 (44.8587)
  IL-6: Day 14 | 15.190 (13.9920) | 60.895 (68.6252) | 3.460 (4.2615) | 16.038 (38.8392)
  IL-6: Day 21 | 3.984 (4.0063) | 50.969 (60.5058) | 4.365 (3.7982) | 14.882 (36.1528)
  IL-6: Day 28: number analyzed (Participants) | 2 | 5 | 8 | 6
  IL-6: Day 28 | 6.569 (6.9839) | 39.678 (74.2068) | 4.413 (7.9900) | 7.208 (16.5226)
  IL-6: Month 2: number analyzed (Participants) | 0 | 2 | 5 | 7
  IL-6: Month 2 |  | 5.774 (8.1652) | 3.650 (2.8818) | 1.317 (1.3573)
  IL-6: Month 3: number analyzed (Participants) | 0 | 1 | 3 | 7
  IL-6: Month 3 |  | 0.000 (NA) — SD was not estimable for a single participant. | 0.924 (1.6003) | 1.489 (1.4878)
  IL-6: Month 4: number analyzed (Participants) | 0 | 1 | 1 | 4
  IL-6: Month 4 |  | 0.000 (NA) — SD was not estimable for a single participant. | 1.501 (NA) — SD was not estimable for a single participant. | 0.473 (0.9450)
  IL-6: Month 6: number analyzed (Participants) | 0 | 1 | 1 | 5
  IL-6: Month 6 |  | 0.000 (NA) — SD was not estimable for a single participant. | 0.000 (NA) — SD was not estimable for a single participant. | 0.954 (0.8722)
  IL-6: Month 9: number analyzed (Participants) | 0 | 0 | 0 | 2
  IL-6: Month 9 |  |  |  | 0.000 (0.0000)
  IL-6: Month 12: number analyzed (Participants) | 0 | 0 | 0 | 1
  IL-6: Month 12 |  |  |  | 0.000 (NA) — SD was not estimable for a single participant.

14. Secondary Outcome: Percentage of Participants With B-cell Aplasia Before and After TAK-007 Administration
Description: B-cell aplasia is defined as <50 B-cells per microliters (µl) of blood.
Time Frame: Pre-dose at Days -5, -4, 0 and post-dose at Days 0, 7, 28 and Months 2, 3, 4, 6, 9, 12
Population: Pharmacodynamic Analysis Set included all participants from the safety analysis set who had a baseline and at least 1 postbaseline sample assessment. Number analyzed is the number of participants with data available for analysis at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 3 | 5 | 10 | 7
percentage of participants
  Pre-dose at Day -5 | 100 | 100 | 70.0 | 71.4
  Pre-dose at Day -4 | 0 | 20.0 | 0 | 0
  Pre-dose at Day 0 | 100 | 100 | 90.0 | 57.1
  Post-dose at 1 hr (+/-15 mins) at Day 0 | 100 | 100 | 90.0 | 85.7
  Post-dose at Day 7 | 100 | 80.0 | 80.0 | 57.1
  Post-dose at Day 28 | 33.3 | 100 | 80.0 | 71.4
  Post-dose at Month 2: number analyzed (Participants) | 0 | 5 | 10 | 7
  Post-dose at Month 2 |  | 40.0 | 50.0 | 71.4
  Post-dose at Month 3: number analyzed (Participants) | 0 | 5 | 10 | 7
  Post-dose at Month 3 |  | 20.0 | 20.0 | 71.4
  Post-dose at Month 4: number analyzed (Participants) | 0 | 5 | 10 | 7
  Post-dose at Month 4 |  | 20.0 | 10.0 | 28.6
  Post-dose at Month 6: number analyzed (Participants) | 0 | 5 | 10 | 7
  Post-dose at Month 6 |  | 20.0 | 10.0 | 42.9
  Post-dose at Month 9: number analyzed (Participants) | 0 | 0 | 0 | 7
  Post-dose at Month 9 |  |  |  | 14.3
  Post-dose at Month 12: number analyzed (Participants) | 0 | 0 | 0 | 7
  Post-dose at Month 12 |  |  |  | 0

15. Secondary Outcome: Percentage of Participants With Detectable Anti-human Leukocyte Antigen (HLA) and Anti-chimeric Antigen Receptor (CAR) Antibodies Before (Prevalence) and After (Incidence) TAK-007 Administration Over Time
Time Frame: Up to 12 months
Population: Safety Analysis Set included all participants who received TAK-007 administration. Number analyzed is the number of participants with data available for analysis at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Dose Escalation: TAK-007 - 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells
Number analyzed (Participants) | 3 | 6 | 10 | 7
percentage of participants
  Anti-HLA Antibodies: Prevalence at Day -5: number analyzed (Participants) | 3 | 5 | 10 | 4
  Anti-HLA Antibodies: Prevalence at Day -5 | 0 | 40.0 | 10.0 | 50.0
  Anti-HLA Antibodies: Prevalence at Day -4: number analyzed (Participants) | 0 | 1 | 0 | 0
  Anti-HLA Antibodies: Prevalence at Day -4 |  | 100 |  |
  Anti-HLA Antibodies: Incidence at Day 14 | 0 | 33.3 | 10.0 | 42.9
  Anti-HLA Antibodies: Incidence at Day 28: number analyzed (Participants) | 2 | 5 | 8 | 7
  Anti-HLA Antibodies: Incidence at Day 28 | 0 | 60.0 | 0 | 42.9
  Anti-HLA Antibodies: Incidence at Month 2: number analyzed (Participants) | 0 | 3 | 5 | 7
  Anti-HLA Antibodies: Incidence at Month 2 |  | 33.3 | 20.0 | 42.9
  Anti-HLA Antibodies: Incidence at Month 3: number analyzed (Participants) | 0 | 2 | 3 | 6
  Anti-HLA Antibodies: Incidence at Month 3 |  | 50.0 | 33.3 | 33.3
  Anti-HLA Antibodies: Incidence at Month 4: number analyzed (Participants) | 0 | 2 | 1 | 4
  Anti-HLA Antibodies: Incidence at Month 4 |  | 50.0 | 0 | 50.0
  Anti-HLA Antibodies: Incidence at Month 6: number analyzed (Participants) | 0 | 1 | 1 | 4
  Anti-HLA Antibodies: Incidence at Month 6 |  | 0 | 0 | 50.0
  Anti-HLA Antibodies: Incidence at Month 9: number analyzed (Participants) | 0 | 1 | 0 | 2
  Anti-HLA Antibodies: Incidence at Month 9 |  | 0 |  | 50.0
  Anti-HLA Antibodies: Incidence at Month 12: number analyzed (Participants) | 0 | 1 | 0 | 1
  Anti-HLA Antibodies: Incidence at Month 12 |  | 100 |  | 0
  Anti-CAR Antibodies: Prevalence at Day -5: number analyzed (Participants) | 3 | 5 | 10 | 6
  Anti-CAR Antibodies: Prevalence at Day -5 | 0 | 0 | 0 | 0
  Anti-CAR Antibodies: Prevalence at Day -4: number analyzed (Participants) | 0 | 0 | 0 | 0
  Anti-CAR Antibodies: Incidence at Day 14 | 0 | 0 | 0 | 0
  Anti-CAR Antibodies: Incidence at Day 28: number analyzed (Participants) | 2 | 6 | 8 | 7
  Anti-CAR Antibodies: Incidence at Day 28 | 0 | 0 | 0 | 0
  Anti-CAR Antibodies: Incidence at Month 2: number analyzed (Participants) | 0 | 3 | 5 | 7
  Anti-CAR Antibodies: Incidence at Month 2 |  | 0 | 0 | 0
  Anti-CAR Antibodies: Incidence at Month 3: number analyzed (Participants) | 0 | 2 | 3 | 7
  Anti-CAR Antibodies: Incidence at Month 3 |  | 0 | 0 | 0
  Anti-CAR Antibodies: Incidence at Month 4: number analyzed (Participants) | 0 | 2 | 1 | 4
  Anti-CAR Antibodies: Incidence at Month 4 |  | 0 | 0 | 0
  Anti-CAR Antibodies: Incidence at Month 6: number analyzed (Participants) | 0 | 1 | 1 | 5
  Anti-CAR Antibodies: Incidence at Month 6 |  | 0 | 0 | 0
  Anti-CAR Antibodies: Incidence at Month 9: number analyzed (Participants) | 0 | 1 | 0 | 2
  Anti-CAR Antibodies: Incidence at Month 9 |  | 0 |  | 0
  Anti-CAR Antibodies: Incidence at Month 12: number analyzed (Participants) | 0 | 1 | 0 | 1
  Anti-CAR Antibodies: Incidence at Month 12 |  | 0 |  | 0

16. Secondary Outcome: Percentage of Participants With Positive Replication Competent Retrovirus (RCR) Test Results Before (Prevalence) and After (Incidence) TAK-007 Administration Over Time
Time Frame: Up to 60 months
Reporting Status: Not Posted, anticipated posting 2039-12

ADVERSE EVENTS:
Time Frame: Up to data cut-off date, 1 July 2024 (up to 31.66 months)
Description: Safety Analysis Set included all participants who received TAK-007 administration.
Groups:
- Dose Escalation: TAK-007: 200×10^6 CD19-CAR+ Viable NK Cells: Participants received lymphodepleting chemotherapy per day IV for 3 days followed by TAK-007 -200×10^6 CD19-CAR+ viable NK cells, single-dose, IV infusion, once on Day 0.
- Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007: Participants with r/r LBCL received lymphodepleting chemotherapy per day IV for 3 days followed by TAK-007 at the dose level(s) selected based on the dose escalation part (800×10^6 CD19-CAR+ viable NK cells), as a single-dose, IV infusion, once on Day 0 to determine RP2D.
- Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007: Participants with r/r iNHL received lymphodepleting chemotherapy per day IV for 3 days followed by TAK-007 at the dose level(s) selected based on the dose escalation part (800×10^6 CD19-CAR+ viable NK cells), as a single-dose, IV infusion, once on Day 0 to determine RP2D.
Arm/Group | Dose Escalation: TAK-007: 200×10^6 CD19-CAR+ Viable NK Cells | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007
All-Cause Mortality (participants affected / at risk) | 2/3 | 3/6 | 5/10 | 0/7
Serious Adverse Events (participants affected / at risk) | 3/3 | 4/6 | 8/10 | 5/7
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 10/10 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: TAK-007: 200×10^6 CD19-CAR+ Viable NK Cells (N=3) | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells (N=6) | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 (N=10) | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 (N=7)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0
High grade B-cell lymphoma refractory (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation: TAK-007: 200×10^6 CD19-CAR+ Viable NK Cells (N=3) | Dose Escalation: TAK-007 - 800×10^6 CD19-CAR+ Viable NK Cells (N=6) | Dose Expansion: Cohort 1 (LBCL 3L+): TAK-007 (N=10) | Dose Expansion: Cohort 2 (iNHL 3L+): TAK-007 (N=7)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 5 | 5 | 2
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Blood fibrinogen decreased (Investigations) | 0 | 1 | 0 | 0
Blood immunoglobulin G decreased (Investigations) | 0 | 0 | 2 | 0
Blood immunoglobulin M decreased (Investigations) | 0 | 0 | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Coronavirus infection (Infections and infestations) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 1 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 3
Disturbance in attention (Nervous system disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 3 | 1
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Enterococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Enterovirus infection (Infections and infestations) | 0 | 1 | 0 | 0
Evans syndrome (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 2 | 2 | 6 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Folate deficiency (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 2 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 1
Hypotension (Vascular disorders) | 2 | 3 | 2 | 1
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0 | 0
Intranasal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 5 | 1
Lymphocyte count increased (Investigations) | 0 | 0 | 1 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 4 | 6 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 5 | 2
Neutrophil count decreased (Investigations) | 1 | 1 | 2 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 2 | 1 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1
Oral mucosal exfoliation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 1 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 1 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Serum ferritin increased (Investigations) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 2 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Vagus nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 6 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT05020015/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT05020015/SAP_001.pdf